CLINICAL TRIAL: NCT01523886
Title: Optimization of Surgical Conditions During Laparoscopic Cholecystectomy With Deep or Moderate Neuromuscular Blockade
Brief Title: The Muscle Relaxation-study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Herlev Hospital (Other)
Responsible Party: Principal Investigator, Anne Kathrine Staehr-Rye, Clinical research assistent, Herlev Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2011-441
Record Dates: First submitted 2012-01-19; First posted 2012-02-01 (Estimated); Results first posted 2014-04-21 (Estimated); Last update posted 2014-04-21 (Estimated); Status verified 2014-03

CONDITIONS: Cholecystectomy, Laparoscopic
MeSH Terms: interventions — Rocuronium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Deep neuromuscular blockade (Active Comparator)
  Interventions: Drug: Rocuronium
- Moderate neuromuscular blockade (Placebo Comparator)
  Interventions: Drug: Rocuronium

INTERVENTIONS:
Drug: Rocuronium — Intravenous use: 0.3 mg/kg before intubation and 0,7 mg after intubation followed by infusion with 0,3-0,4 mg/kg/h
  Other Names: Esmeron
  Arms: Deep neuromuscular blockade
Drug: Rocuronium — Intravenous use: 0,3 mg/kg followed by NaCl-infusion
  Other Names: Esmeron
  Arms: Moderate neuromuscular blockade

SUMMARY:
The purpose of this investigation is to compare the surgical conditions during laparoscopic cholecystectomy at a low intra-abdominal pressure with deep or moderate muscle relaxation.

The primary hypothesis is that surgical conditions during laparoscopic cholecystectomy are better with deep muscle relaxation than moderate muscle relaxation.

DETAILED DESCRIPTION:
The purpose of this investigation is to compare the surgical conditions with two degrees of neuromuscular blockade in patients who have laparoscopic cholecystectomy done with pneumoperitoneum 8 mmHg.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years
* Scheduled for elective laparoscopic cholecystectomy
* Can read and understand danish
* Women must be post-menopausal, sterilized or use safe contraception in the form of a coil or oral anti-contraceptives

Exclusion Criteria:

* Known allergy to medications that are included in the project
* Presence of severe renal disease, neuromuscular disease, reduced liver function
* Nursing or pregnant
* Indication for crash induction
* For fertile women: Missing negative pregnancy-test

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2012-03; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne K Staehr, MD, Principal Investigator — Department of anesthesia, Herlev Hospital, Denmark; Mona R Gätke, MD, Ph.D, Study Chair — Department of anesthesia, Herlev Hospital
Locations (1):
- Department of anesthesia and department of gastro-intestinale diseases, Aleris-Hamlet, Soeborg, Denmark

REFERENCES:
- [Derived] Staehr-Rye AK, Rasmussen LS, Rosenberg J, Juul P, Gatke MR. Optimized surgical space during low-pressure laparoscopy with deep neuromuscular blockade. Dan Med J. 2013 Feb;60(2):A4579. PMID 23461992

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Deep Neuromuscular Blockade | Moderate Neuromuscular Blockade
Started | 25 | 24
Completed | 25 | 23
Not Completed | 0 | 1
Not completed — surgery cancelled | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Deep Neuromuscular Blockade | Moderate Neuromuscular Blockade | Total
Number analyzed (Participants) | 25 | 23 | 48
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 45 [42 to 49] | 48 [35 to 59] | 45 [36 to 56]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 17 | 32
  Male | 10 | 6 | 16
Region of Enrollment [Number; unit: participants]
  Denmark | 25 | 23 | 48

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Patients With Optimal Surgical Space Conditions ( 1 at a 4-step Scale) Assessed at the Time During Surgery, When View Was Less
Description: The surgical space conditions (4-stage scale) assessed at the time during surgery, when view was less. The laparoscopies were performed by experienced surgeons, whom were asked to evaluate surgical space conditions with a 4-point scale : Grade 1 ("optimal") = "optimal" surgical space conditions; Grade 2 (good) = non-optimal conditions, but an intervention was not considered; Grade 3 (acceptable) = an intervention was considered in order to improve surgical space; Grade 4 (poor) = inadequate conditions and an intervention was necessary in order to ensure acceptable surgical space.
Time Frame: From surgical incision to last suture has been placed, an expected average of 30 minutes
Measure: Number; unit: percentage of patients
Arm/Group | Deep Neuromuscular Blockade | Moderate Neuromuscular Blockade
Number analyzed (Participants) | 25 | 23
percentage of patients | 28 | 4

2. Secondary Outcome: Surgical Space Conditions
Description: The surgical space conditions (VAS 0-100) assessed at the time during surgery, when they were poorest
Time Frame: From surgical incision to last suture has been placed, an expected average of 30 minutes.
Reporting Status: Not Posted

3. Secondary Outcome: Surgical Space Conditions
Description: The average surgical space conditions (VAS 0-100 and 4-stage scale) during the procedure.
Time Frame: From surgical incision to last suture has been placed, an expected average of 30 minutes.
Reporting Status: Not Posted

4. Secondary Outcome: Surgical Space Conditions
Description: The surgical space conditions during dissection of the gallbladder (4-stage scale and VAS 0-100).
Time Frame: During dissection of the gallbladder
Reporting Status: Not Posted

5. Secondary Outcome: Pain
Description: Pain (shoulder, incision, deep abdominal and general) as the area under the curve from preoperatively to 7 days after surgery.
Time Frame: Preoperatively to 7 days after surgery
Reporting Status: Not Posted

6. Secondary Outcome: Pain
Description: Pain (shoulder, incision, deeop abdominal and general) at arrival to the postanesthesia care department, 2 hours and 1 day after surgery.
Time Frame: At arrival to the postanesthesia care department, 2 hours and 1 day after surgery
Reporting Status: Not Posted

7. Secondary Outcome: Normal Functional Level
Description: Numer of days before re-establing normal functional level
Time Frame: from the day of surgery to re-establishing normal functional level - an expected average of 7 days.
Reporting Status: Not Posted

8. Secondary Outcome: Surgical Procedures at Low Pneumoperitoneum
Description: Number of procedures which can be done with pneumoperitoneum 8 mmHg
Time Frame: From surgical incision to last suture has been placed, an expected average of 30 minutes.
Reporting Status: Not Posted

9. Secondary Outcome: Duration of Surgery
Description: Duration of surgery
Time Frame: From surgical incision to last suture has been placed.
Reporting Status: Not Posted

10. Secondary Outcome: Duration of Anesthesia
Description: Duration of anesthesia
Time Frame: From induction of anesthesia to patient ready to leave the operating theatre
Reporting Status: Not Posted

11. Secondary Outcome: Consumption of Analgesics
Description: Consumption of analgesics during the first 24 hours after surgery
Time Frame: The first 24 hours after surgery
Reporting Status: Not Posted

12. Secondary Outcome: Nausea and Vomiting
Description: The incidence of nausea and vomiting during the first 24 hours after surgery
Time Frame: The first 24 hours after surgery
Reporting Status: Not Posted

13. Secondary Outcome: Anti-emetics
Description: Use of anti-emetics during the first 24 hours after surgery
Time Frame: During the first 24 hours after surgery
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Deep Neuromuscular Blockade | Moderate Neuromuscular Blockade
Serious Adverse Events (participants affected / at risk) | 3/25 | 1/23
Other Adverse Events (participants affected / at risk) | 12/25 | 11/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Deep Neuromuscular Blockade (N=25) | Moderate Neuromuscular Blockade (N=23)
Prolonged hospitalization (Surgical and medical procedures) | 1 (1) | 1 (1) — Postoperative observation
Readmission to hospital (Surgical and medical procedures) | 2 (2) | 0 (0) — Undiagnosed gallstones in the common bile duct
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Deep Neuromuscular Blockade (N=25) | Moderate Neuromuscular Blockade (N=23)
Pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1)
Pain (Surgical and medical procedures) | 4 (4) | 6 (6)
Headache and vertigo (Surgical and medical procedures) | 3 (3) | 3 (3)
Bleeding from sutur (Surgical and medical procedures) | 0 (0) | 1 (1)
hoarseness (Gastrointestinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No